CLINICAL TRIAL: NCT00783185
Title: Dual Diagnosis Psychosis and Substance Abuse: Short- and Middle-term Changes in Symptomatology After Visiting a Group Education Programme to Reduce Consumption of Cannabis
Brief Title: Dual Diagnosis (Psychosis and Cannabismisuse): Comparison of Specialized Treatment Versus Unspecified Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Hans Watzl, Dr., University of Konstanz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRET
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2008-10

CONDITIONS: Psychotic Disorders; Marijuana Abuse; Intervention
Keywords: psychotic disorders; cannabis; intervention
MeSH Terms: conditions — Psychotic Disorders; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT (Experimental): Anti-Cannabis-Consumption-Training
  Interventions: Behavioral: Cannabis-Consumption-Reduction-Training
- CG (Active Comparator): Control group
  Interventions: Behavioral: Social competence Training

INTERVENTIONS:
Behavioral: Cannabis-Consumption-Reduction-Training — 8 sessions within 4 weeks (twice a week, 45 minutes each) Cognitive behavioral therapy with focus on cannabis abuse
  Arms: ACT
Behavioral: Social competence Training — 8 sessions within 4 weeks (twice a week, 45 minutes) training to develop and ameliorate social competences
  Arms: CG

SUMMARY:
Intention of the study is to examine, if the symptomatology of dual diagnosis patients is less severe after a special indication training for reduction of cannabis consumption in comparison to unspecified trainings.

Point of interest is psychopathology and consumerism.

DETAILED DESCRIPTION:
Dual diagnosis patients (psychosis and cannabis abuse) account for more clinical admissions than single diagnosis patients.

Cannabis misuse is a known risk factor for recurrence of psychosis.

A specified intervention on the basis of a manual for schizophrenic substance abusers is administered to inpatients in a specialized unit for young schizophrenic patients in a psychiatric hospital.

The control group, same indication (psychotic disorder and cannabis misuse) receives social competence training (specified for schizophrenic patients as well).

Admission to groups is randomly.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia and disorders with psychotic features
* Misuse of cannabis during 12 months preceding admission to hospital

Exclusion Criteria:

* Not able to attend training twice a week for 45 minutes (concentration, attention, psychotic symptoms, agitation)
* Discharge from hospital before completion of training

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
PANSS Positive and Negative Symptom Scale | post intervention, six months follow-up

SECONDARY OUTCOMES:
Urinstatus for cannabinoids | weekly during and post intervention, follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hans Watzl, Dr., Principal Investigator — University of Konstanz
Locations (1):
- University of Konstanz, Konstanz, Baden-Wurttemberg, Germany